CLINICAL TRIAL: NCT03646578
Title: Maternal Anxiety Related to How the Pediatrician Provided Prenatal Information About Preterm Birth
Acronym: Infoprema
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0038
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Preterm Birth
Keywords: maternal anxiety
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: State of anxiety — Patient anxiety assessment by STAI-Y-A self-assessment questionnaire provided before and after pediatric interview.
  The assessment is given to patients upon arrival in the hospitalization service of pregnancies and again after the pediatric interview. This pediatric interview should take place between 1 and 7 days after admission to the hospital ward.The second part includes a 6-week inclusion period with assessment of patients' state of anxiety by a STAI-Y-A self-assessment questionnaire given before and after pediatric interview associated with the delivery of a written document. on prematurity.

SUMMARY:
Women hospitalized for preterm labor require clear information about prematurity.

This study assessed whether or not specific written information about prematurity delivered at admission to the unit combined with an oral explanation from a pediatrician would decrease women's anxiety compared to an oral explanation alone. This was a prospective, single-center observational study.Women were included in the high-risk pregnancies department and distributed into two groups: receiving ''only oral'' information for a prenatal clinical consultation with a senior pediatrician or receiving ''combined'' oral information + a booklet about prematurity given to the women at admission. The primary endpoint was the change in anxiety-state (before and after the information procedure) evaluated by the State Trait Anxiety Inventory-Y (STAI-Y).

DETAILED DESCRIPTION:
Women hospitalized for preterm labor require clear information about prematurity.

This study assessed whether or not specific written information about prematurity delivered at admission to the unit combined with an oral explanation from a pediatrician would decrease women's anxiety compared to an oral explanation alone. Material and methods.This was a prospective, single-center observational study.Women were included in the high-risk pregnancies department and distributed into two groups: receiving ''only oral'' information for a prenatal clinical consultation with a senior pediatrician or receiving ''combined'' oral information

+ a booklet about prematurity given to the women at admission.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in the service of pregnancies and having a risk of premature delivery.
* Term <34 SA

Exclusion Criteria:

* Term ≥ 34 SA
* no understanding of the questionnaire
* foetus presenting a pathology or malformation that is life-threatening
* patient presenting a risk of delivery before passing the pediatrician or presenting a risk of imminent delivery
* patient hospitalized without risk of premature delivery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 60 hospitalized patients at risk of preterm birth
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Mesure of the State of anxiety of patients with a risk of premature delivery | 3months
  The objective of the study is to evaluate the impact of the written medical information about prematurity delivered at admission to the unit by the doctor, on the state of anxiety of patients hospitalized with a risk of premature delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Tourneux, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No